CLINICAL TRIAL: NCT00397163
Title: A Clinical Study Investigating Ischemic Preconditioning in Type II Diabetic Patients Undergoing Coronary Artery Bypass Graft Surgery.
Brief Title: Effect of Remote Ischemic Preconditioning in Patient Undergoing Cardiac Bypass Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University College London Hospitals (Other)
Responsible Party: Principal Investigator, Derek Yellon, Director of the Hatter Cardiovascular Institute, University College London Hospitals
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 01/0128
Record Dates: First submitted 2006-11-06; First posted 2006-11-08 (Estimated); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Coronary Heart Disease
Keywords: Coronary artery bypass graft surgery; Remote ischemic preconditioning; Troponin-T
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Remote preconditioning (Active Comparator): Simultaneous inflation (5min) and deflation (5min) of cuffs placed on upper arm and thigh - cycle repeated 2 times
  Interventions: Procedure: Remote ischemic preconditioning
- Placebo (Placebo Comparator): Deflated cuffs placed on upperarm and thigh for 20 minutes
  Interventions: Procedure: Placebo

INTERVENTIONS:
Procedure: Remote ischemic preconditioning — Blood pressure cuff inflation
  Other Names: Remote Ischaemic Preconditioning
  Arms: Remote preconditioning
Procedure: Placebo — Deflated cuff on upper arm and thigh for 20 min
  Other Names: Control
  Arms: Placebo

SUMMARY:
During coronary artery bypass graft surgery, injury occurs to the heart muscle. Some of this injury is due to the deprivation of oxygen and nutrients to the heart (a process called ischemia) during the surgery itself. The objective of this study is to examine whether remote ischaemic preconditioning (RIPC), in which the application of transient ischemia to the forearm and thigh (through the inflation of blood pressure cuffs placed on the right upper arm and upper thigh) may reduce the injury to the heart muscle sustained during cardiac surgery.

The study hypothesis is: remote ischemic preconditioning will protect the heart and improve short-term clinical outcomes during coronary artery bypass graft surgery.

DETAILED DESCRIPTION:
Ischemic heart disease (IHD) is currently the leading cause of morbidity and mortality in the developed world, and is set to become the leading cause of death in the world by the year 2020, according to the World Health Organisation. Patients with severe IHD that require coronary artery bypass graft (CABG) surgery, although protected by techniques such as cross-clamp fibrillation and cardioplegia, still sustain significant myocardial injury as evidenced by perioperative troponin T or I or CK-MB release. Novel treatment strategies are required to limit the myocardial injury sustained by patients undergoing CABG surgery in order to improve the clinical outcomes of this patient group.

One such cardioprotective strategy is remote ischemic preconditioning(RIPC) which describes the cardioprotection obtained from inducing ischemia in tissue or an organ remote from the heart. Our laboratory and others have established RIPC using forearm ischemia (induced by an automated cuff applied to the upper arm) as an effective cardioprotective intervention in children undergoing corrective cardiac surgery for congenital heart disease and in adults undergoing CABG surgery. In this study we investigate whether simultaneous inflation/deflation of cuffs placed on the upper arm and thigh can reduce peri-operative myocardial injury and improve short-term outcomes in patients undergoing CABG surgery.

Eligible patients will be those patients undergoing elective CABG surgery who are >18 years old, with no significant renal or hepatic disease, and have not had a recent AMI (within 1 month).

Consented patients will randomized to RIPC treatment or control.The RIPC protocol will comprise simultaneous 2 x 5 minutes of forearm and lower leg ischemia (with an automated pressure cuff inflated to 200 mmHg) with an intervening 5 minutes of reperfusion (during which the cuff is deflated) between each inflation. The control protocol will comprise a deflated cuff being placed on the upper arm and thigh for 20 minutes. The RIPC protocol will be implemented after the patients have been anesthetized and immediately prior to CABG surgery.

The measured endpoint of cardioprotection will be troponin-T release at 0, 12, 24, 48 and 72 hours following CABG surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing elective CABG surgery

Exclusion Criteria:

* <18 years old
* Significant renal or hepatic disease
* Previous acute myocardial infarction (within 4 weeks)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2010-12 (Actual); Primary Completion 2017-01-13 (Actual); Study Completion 2017-01-13 (Actual)

PRIMARY OUTCOMES:
Troponin-T release over the perioperative 72-hour period. | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Derek M Yellon, PhD DSc, Principal Investigator — The Hatter Cardiovascular Institute, UCL.
Locations (1):
- The UCLH Heart Hospital, 14-16 Westmoreland St., London, United Kingdom

REFERENCES:
- [Background] Kharbanda RK, Li J, Konstantinov IE, Cheung MM, White PA, Frndova H, Stokoe J, Cox P, Vogel M, Van Arsdell G, MacAllister R, Redington AN. Remote ischaemic preconditioning protects against cardiopulmonary bypass-induced tissue injury: a preclinical study. Heart. 2006 Oct;92(10):1506-11. doi: 10.1136/hrt.2004.042366. Epub 2006 Jul 3. PMID 16818489
- [Background] Loukogeorgakis SP, Panagiotidou AT, Broadhead MW, Donald A, Deanfield JE, MacAllister RJ. Remote ischemic preconditioning provides early and late protection against endothelial ischemia-reperfusion injury in humans: role of the autonomic nervous system. J Am Coll Cardiol. 2005 Aug 2;46(3):450-6. doi: 10.1016/j.jacc.2005.04.044. PMID 16053957
- [Background] Broadhead MW, Kharbanda RK, Peters MJ, MacAllister RJ. KATP channel activation induces ischemic preconditioning of the endothelium in humans in vivo. Circulation. 2004 Oct 12;110(15):2077-82. doi: 10.1161/01.CIR.0000144304.91010.F0. Epub 2004 Oct 4. PMID 15466634
- [Background] Kharbanda RK, Mortensen UM, White PA, Kristiansen SB, Schmidt MR, Hoschtitzky JA, Vogel M, Sorensen K, Redington AN, MacAllister R. Transient limb ischemia induces remote ischemic preconditioning in vivo. Circulation. 2002 Dec 3;106(23):2881-3. doi: 10.1161/01.cir.0000043806.51912.9b. PMID 12460865
- [Background] Kharbanda RK, Peters M, Walton B, Kattenhorn M, Mullen M, Klein N, Vallance P, Deanfield J, MacAllister R. Ischemic preconditioning prevents endothelial injury and systemic neutrophil activation during ischemia-reperfusion in humans in vivo. Circulation. 2001 Mar 27;103(12):1624-30. doi: 10.1161/01.cir.103.12.1624. PMID 11273988
- [Background] Cheung MM, Kharbanda RK, Konstantinov IE, Shimizu M, Frndova H, Li J, Holtby HM, Cox PN, Smallhorn JF, Van Arsdell GS, Redington AN. Randomized controlled trial of the effects of remote ischemic preconditioning on children undergoing cardiac surgery: first clinical application in humans. J Am Coll Cardiol. 2006 Jun 6;47(11):2277-82. doi: 10.1016/j.jacc.2006.01.066. Epub 2006 May 15. PMID 16750696
- [Background] Konstantinov IE, Li J, Cheung MM, Shimizu M, Stokoe J, Kharbanda RK, Redington AN. Remote ischemic preconditioning of the recipient reduces myocardial ischemia-reperfusion injury of the denervated donor heart via a Katp channel-dependent mechanism. Transplantation. 2005 Jun 27;79(12):1691-5. doi: 10.1097/01.tp.0000159137.76400.5d. PMID 15973170
- [Background] Kristiansen SB, Henning O, Kharbanda RK, Nielsen-Kudsk JE, Schmidt MR, Redington AN, Nielsen TT, Botker HE. Remote preconditioning reduces ischemic injury in the explanted heart by a KATP channel-dependent mechanism. Am J Physiol Heart Circ Physiol. 2005 Mar;288(3):H1252-6. doi: 10.1152/ajpheart.00207.2004. Epub 2004 Oct 21. PMID 15498829
- [Background] Konstantinov IE, Arab S, Kharbanda RK, Li J, Cheung MM, Cherepanov V, Downey GP, Liu PP, Cukerman E, Coles JG, Redington AN. The remote ischemic preconditioning stimulus modifies inflammatory gene expression in humans. Physiol Genomics. 2004 Sep 16;19(1):143-50. doi: 10.1152/physiolgenomics.00046.2004. Epub 2004 Aug 10. PMID 15304621
- [Derived] Candilio L, Malik A, Ariti C, Barnard M, Di Salvo C, Lawrence D, Hayward M, Yap J, Roberts N, Sheikh A, Kolvekar S, Hausenloy DJ, Yellon DM. Effect of remote ischaemic preconditioning on clinical outcomes in patients undergoing cardiac bypass surgery: a randomised controlled clinical trial. Heart. 2015 Feb;101(3):185-92. doi: 10.1136/heartjnl-2014-306178. Epub 2014 Sep 24. PMID 25252696
- [Derived] Venugopal V, Hausenloy DJ, Ludman A, Di Salvo C, Kolvekar S, Yap J, Lawrence D, Bognolo J, Yellon DM. Remote ischaemic preconditioning reduces myocardial injury in patients undergoing cardiac surgery with cold-blood cardioplegia: a randomised controlled trial. Heart. 2009 Oct;95(19):1567-71. doi: 10.1136/hrt.2008.155770. Epub 2009 Jun 8. PMID 19508973
- [Derived] Hausenloy DJ, Mwamure PK, Venugopal V, Harris J, Barnard M, Grundy E, Ashley E, Vichare S, Di Salvo C, Kolvekar S, Hayward M, Keogh B, MacAllister RJ, Yellon DM. Effect of remote ischaemic preconditioning on myocardial injury in patients undergoing coronary artery bypass graft surgery: a randomised controlled trial. Lancet. 2007 Aug 18;370(9587):575-9. doi: 10.1016/S0140-6736(07)61296-3. PMID 17707752